CLINICAL TRIAL: NCT07237724
Title: Effects of Motor Imagery on Pain, Function, Endurance, Kinesiophobia and Sleep Quality in Patients With Non-specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Sara Hamdi Mohamed Kamal Shalabi, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/020-65
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Non-specific Low Back Pain
Keywords: action observation; Non-specific Low Back Pain; core exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Exercise Program (Active Comparator): Participants receive supervised core exercise therapy 3 times per week for 6 weeks.
  Interventions: Other: Core Exercise Program
- Core Exercise + Action Observation (Experimental): Participants receive the same core exercise therapy plus an action observation session before each treatment.
  Interventions: Other: Action Observation Therapy

INTERVENTIONS:
Other: Core Exercise Program — * The patients will do their exercises at the clinic as face to face sessions. All sessions will be conducted under the supervision of a physiotherapist
  * patients will receive core exercises program, 3 days per week
  * Treatment duration is 6 weeks
  Arms: Core Exercise Program
Other: Action Observation Therapy — * The patients will do their exercises at the clinic as face to face sessions. All sessions will be conducted under the supervision of a physiotherapist
  * patients will receive the same core exercises program as the Active comparator group, 3 days per week for 6 weeks
  * This group will receive action observation therapy for 6 minutes before every exercise therapy session. they will watch videos of 2 different activates, the duration of each video is 3 minutes and will be recorded from 3 planes (front, back and lateral )
  Arms: Core Exercise + Action Observation

SUMMARY:
Non-specific low back pain (NSLBP) is one of the most common musculoskeletal disorders all over the world and a leading cause of disability. It affects individuals across different age groups and is typically characterized by pain, stiffness, and functional limitations that reduce physical activity and overall quality of life. Among established clinical approaches, Core exercises are frequently used in the management of LBP, reducing pain and improving functionality by stabilizing the spine. However, despite their widespread use, there is limited evidence on the effectiveness of combining core exercises with cognitive interventions, such as action observation.

Motor imagery (MI) and action observation (AO) offer practical, low-cost approaches that can be easily integrated into rehabilitation programs. Motor imagery involves the individual visualizing the physical movement in their mind without performing it, while action observation involves learning specific movements by observing them. These techniques can strengthen the effectiveness of physical exercises by increasing neuromuscular activation. However, it has been reported that motor imagery-based cortical processes facilitate the reorganization of sensory-motor functions during daily activities in LBP patients. Studies in this area are quite limited. The effectiveness of action observation therapy, which is primarily effective in neurological conditions, has not been investigated in non-specific low back pain. Therefore, in this study, the effects of combining action observation therapy with a core exercise program, Pain, Function, Endurance, Kinesiophobia, and Sleep Quality in patients with non-specific low back pain will be examined.

The study aims to investigate the effects of combining action observation therapy with core exercises compared with core exercises alone in patients with NSLBP. Patients attending Fizyowell physiotherapy and Healthy Services clinic who meet the inclusion criteria will be included in the study. This study seeks to explore the potential benefits of integrating cognitive techniques into a conventional exercise-based rehabilitation for NSLBP.

To establish participant eligibility before the study begins, a standardized demographic data form will be collected from all subjects who volunteered to participate in the study, including gender, age, height, weight, education, marital status, chronic diseases and medication use, smoking, and alcohol use. In addition, the Mini-Mental State Examination (MMSE) will be used to assess the patient's mental state, determine the ability to understand and follow instructions, and identify cognitive disorders that may make it difficult to perform mental interventions. The Movement Imagery Questionnaire-3 (MIQ-3) will be used to determine each participant's motor imagery ability. Once eligibility is confirmed, baseline assessments will be conducted, including pain intensity measured by the Visual Analog Scale (VAS), functional disability assessed using the Oswestry Low Back Pain Disability Index Questionnaire, kinesiophobia evaluated with the Tampa Scale for Kinesiophobia (TSK), core endurance tested through standardized endurance measures, and sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI).

After the initial evaluation, the treatment program will be started. Advances in the treatment method specific to the groups they belong to are explained in detail below.

Treatment:

After the first evaluation, the core exercise program will be applied to the patients in Group 1, 3 days per week for 6 weeks. All sessions will be conducted under the supervision of a physiotherapist at the clinic.

Group 2: Conservative Treatment + Action Observation Program. This group will have action observation therapy in addition to the core exercise program. The patients in this group will receive an action observation therapy for 6 minutes before each exercise therapy session. They will watch videos of 2 different activities, the duration of each video is 3 minutes, and they were recorded from 3 planes (frontal, back, and lateral).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Being a volunteer.
* Having nonspecific chronic low back pain for three months or more.
* No obvious structural or anatomical abnormality that could explain the pain.
* Scoring 24 or more out of 30 on the Mini-Mental State Examination.
* Those who score high in terms of imagery ability on the MIQ-3 questionnaire.
* Not having any pathology in vision or hearing

Exclusion Criteria:

* pregnancy
* Having a painful spinal deformity.
* Having a spinal surgery
* Having a mental illness and/or communication problem.
* Having pain radiating to the lower extremity.
* Having any back disease diagnosed by a specialist physician other than non-specific chronic back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Baseline (Day 1) and After 6 Weeks of Treatment
  The Visual Analog Scale (VAS) is an important instrument used for measuring the severity of low back pain at rest and during physical activity. It provides a simple, validated method of transforming subjective pain experiences into numerical values suitable for statistical analysis. Participants will be asked to rate their pain intensity on a scale from 0 to 10, where 0 represents "no pain" and 10 represents "unbearably severe pain".

SECONDARY OUTCOMES:
Functionality Level | Baseline (Day 1) and Week 6.
  Oswestry Low Back Pain Disability Index Questionnaire (ODI) The Oswestry Questionnaire is a widely used tool to assess the level of functional disability in patients with low back pain. It consists of 10 sections: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and degree of pain change. Each section has 6 response options scored from 0 to 5, with higher scores indicating greater disability. The total score ranges from 0 to 50, which may be converted to a percentage (0-100% disability). A higher total score reflects a higher level of functional disability.
Core Muscle Endurance | At baseline and after 6 weeks of intervention
  Trunk Flexor Test - Trunk Extensor Test -Side Bridge Test - Prone plank Test
Kinesiofobia Level | Baseline and Week 6.
  "Kinesiophobia" is a term referring to the fear of movement and physical activity due to fear of reinjury, pain or the belief that any physical effort may lead to further harm or complications. The Tampa Scale for Kinesiophobia (TSK) is a validated 17-item questionnaire used to assess the fear of movement and reinjury. Each item is scored from 1 (strongly disagree) to 4 (strongly agree), producing a total score range of 17 to 68. Higher scores indicate greater fear of movement (higher kinesiophobia).
Sleep Quality | From the start of treatment until 6 week after the end of treatment
  Pittsburgh Sleep Quality Index (PSQI):
  The Pittsburgh Sleep Quality Index is a validated 19-item self-report questionnaire assessing sleep quality over the past month. It produces a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Hamdi Shalabi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy considerations and restrictions imposed by the ethics committee

REFERENCES:
- [Result] Salik Sengul Y, Kaya N, Yalcinkaya G, Kirmizi M, Kalemci O. The effects of the addition of motor imagery to home exercises on pain, disability and psychosocial parameters in patients undergoing lumbar spinal surgery: A randomized controlled trial. Explore (NY). 2021 Jul-Aug;17(4):334-339. doi: 10.1016/j.explore.2020.02.001. Epub 2020 Feb 22. PMID 32147444
- [Result] Ozturk O, Bombaci H, Kececi T, Algun ZC. Effects of additional action observation to an exercise program in patients with chronic pain due to knee osteoarthritis: A randomized-controlled trial. Musculoskelet Sci Pract. 2021 Apr;52:102334. doi: 10.1016/j.msksp.2021.102334. Epub 2021 Jan 24. PMID 33582621
- [Result] Salik Sengul Y, Yilmaz A, Kirmizi M, Kahraman T, Kalemci O. Effects of stabilization exercises on disability, pain, and core stability in patients with non-specific low back pain: A randomized controlled trial. Work. 2021;70(1):99-107. doi: 10.3233/WOR-213557. PMID 34487008